CLINICAL TRIAL: NCT04962906
Title: Randomised Phase II Study to Evaluate the Immunogenicity and Safety of Heterologous SARS-CoV-2 Vaccine Schemes (rAd26-rAd5, ChAdOx1 nCoV-19 and BBIBP-CorV).
Brief Title: Study to Evaluate the Immunogenicity and Safety of Heterologous SARS-CoV-2 Vaccine Schemes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ministerio de Salud de Ciudad Autónoma de Buenos Aires (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5143
Record Dates: First submitted 2021-07-08; First posted 2021-07-15 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Vaccines
Keywords: COVID-19 Serological Testing
MeSH Terms: interventions — Gam-COVID-Vac vaccine; ChAdOx1 nCoV-19; BIBP COVID-19 vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All personnel involved in antibody determination shall remain blinded to the assigned strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gam-COVID-Vac / Gam-COVID-Vac (Active Comparator)
  Interventions: Drug: Gam-COVID-Vac / Gam-COVID-Vac
- Gam-COVID-Vac / ChAdOx1 nCoV-19 (Active Comparator)
  Interventions: Drug: Gam-COVID-Vac / Gam-COVID-Vac
- Gam-COVID-Vac / BBIBP-CorV (Active Comparator)
  Interventions: Drug: Gam-COVID-Vac / Gam-COVID-Vac

INTERVENTIONS:
Drug: Gam-COVID-Vac / Gam-COVID-Vac — A comparison of antibody levels against protein S will be performed using the Gam-COVID-Vac / Gam-COVID-Vac group as a control group and the Gam-COVID-Vac / ChAdOx1 nCoV-19 and Gam-COVID-Vac / BBIBP-CorV groups as comparators.
  Other Names: Gam-COVID-Vac / ChAdOx1 nCoV-19; Gam-COVID-Vac / BBIBP-CorV

SUMMARY:
To determine whether a heterologous vaccination regimen in individuals with no known previous history of COVID-19 is non-inferior to that observed with counterpart regimens currently in use in Argentina.

DETAILED DESCRIPTION:
The Covid-19 disease caused by the SARS-COV 2 virus has caused a pandemic with more than 180 million cases worldwide and more than 4 million deaths. In Argentina, this pandemic has had a significant impact, with about 4.5 million cases and about 95,000 deaths. In no more than nine months, medical science developed different vaccines to prevent new cases and mitigate this pandemic.

At the time of the presentation of this research protocol, there are four vaccines for the prevention of COVID-19 approved for emergency use by the National Administration of Medicines, Food and Medical Technology (ANMAT). Of these, three (1-3) are currently available and are part of the vaccination campaign. Of these three vaccines, two use a non-replicating viral vector platform (Gam-COVID-Vac and ChAdOx1 nCoV-19) while one uses an inactivated virus platform (BBIBP-CorV). All require the administration of two doses with an administration interval of at least 21 days.

All these vaccines were designed to be used with a homologous two-dose regimen. However, for both logistical and biomedical reasons, the need to use vaccines in heterologous regimens (one dose of one vaccine and a second dose of another vaccine) is emerging worldwide. The efficacy and safety of this type of regimen has not yet been demonstrated.

In Argentina, there are a large number of people who currently have one dose of Gam-COVID-Vac vaccine and who - even after a period of ≥21 days - have not received the second component. At the same time, the provision of the second component of the Gam-COVID-Vac vaccine is delayed due to production and distribution logistics.

As of June 2021, among the universe of people vaccinated with Gam-COVID, residents of CABA, vaccinated in establishments in the City of Buenos Aires - and excluding deceased and infected people - there were a total of 325,788 people with one dose and ≥22 and ≤90 days since the first dose was administered. In a context of high viral circulation, it is desirable to try to vaccinate as much of the population as possible with a full schedule in the shortest possible time. In addition, new variants of SARS-COV2 virus possessing the E384K genomic variant such as the gamma strain (formerly Manaus), the beta strain (known as South African) and the Delta strain (also known as Indian) have the ability to evade the immune system and therefore most laboratories that have developed vaccines recognise that the efficacy of the vaccines requires two doses.

The use of heterologous schedules is a source of active research in various parts of the world (4-6). However, most of this research is testing the combination of a combination schedule that includes an mRNA vaccine. There is an ongoing study sponsored by the Gamaleya Institute and AstraZeneca that is evaluating the immunogenicity of a scheme similar to the one proposed in this trial. Results from this joint trial would not be available until mid-October (7). No trials have evaluated the combination of rAd26-rAd5 and BBIBP-CorV.

This study will attempt to determine whether administration of a heterologous regimen combining a first dose of Gam-COVID-Vac with a second dose of ChAdOx1 nCoV-19 or BBIBP-CorV results in non-inferior immunogenicity to the homologous regimen used.

The present protocol is therefore oriented to respond to a practical management need and to guarantee the best possible protection to the population through two doses, which is what is considered worldwide as "complete vaccination" according to WHO for the vaccines used by Argentina. The proposed protocol is a pragmatic and public health oriented clinical trial, whose primary objective is to establish whether there are indicators that allow the implementation of a heterologous vaccination scheme. For this, a surrogate endpoint will be used, which is immunogenicity measured by the presence of antibodies against protein S. In addition, the safety of the combination will be evaluated in terms of monitoring self-reported and non-self-reported clinical events by patients.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have received a dose of Gam-COVID-Vac more than 30 days and less than 90 days ago.
* Age between 21 and 65 years.
* Both genders.
* Who have voluntarily agreed to participate in the clinical trial and have provided informed consent.

Exclusion Criteria:

* Known history of COVID in the 6 months prior to study inclusion.
* Known or suspected immunocompromised status by the study investigator for any cause.
* Use of oral or parenteral corticosteroids in the last 30 days.
* Known history of allergy to any vaccine.
* History of anaphylaxis.
* Pregnant or lactating women.
* Known history of autoimmune diseases.
* Persons under treatment for any neoplastic disease within the last 6 months.
* Any serious illness or condition at the discretion of the study investigator (including but not limited to the presence of chronic obstructive pulmonary disease, heart failure, poorly controlled hypertension, poorly controlled diabetes, renal failure).
* Planned medical procedures within two months of randomisation.
* Previous vaccination within the last 30 days with any vaccine.
* Known participation in an ongoing clinical trial.
* Ongoing acute illness.
* Fever (≥37.8 C) at the time of randomisation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
ELISA assessment of IgG anti Spike (UI/ml) | 28 days
  To determine whether a heterologous vaccination regimen in individuals with no known previous history of COVID-19 is non-inferior to that observed with currently used counterpart regimens.
  The determination of the antibody concentration in each of the study arms will be assessed by measuring the IgG antibody concentration using ELISA expressed in IU/ml.
Serious adverse events Adverse events of special interest | 28 days
  To report the combine and specific rate of serious adverse defined as death for any reason, any life-threatening event or any event that require inpatient hospitalization.

SECONDARY OUTCOMES:
Neutralising antibodies against SARS-CoV-2 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ministerio de Salud de la Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No